CLINICAL TRIAL: NCT00222183
Title: Evaluation of the Therapeutic Effect and Local Tolerability of Elidel® Cream 1% (Pimecrolimus) in Chronic Discoid Lupus Erythematosus (dLE) or Subacute Cutaneous Lupus Erythematosus (scLE)
Brief Title: Cutaneous Lupus Erythematosus and Elidel
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Head of the study has left the institution. Study never started.
Sponsor: University of Leipzig (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM-DE-08
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2007-02

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid
Keywords: Lupus erythematodes; Elidel; Pimecrolimus; Chronic discoid lupus erythematosus (dLE); subacute cutaneous lupus erythematosus (scLE)
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid | interventions — pimecrolimus

INTERVENTIONS:
Drug: Elidel (pimecrolimus)

SUMMARY:
This trial evaluates the therapeutic effect of Elidel (pimecrolimus) in comparison to the corresponding vehicle in patients with chronic discoid lupus erythematosus (dLE) or subacute cutaneous lupus erythematosus (scLE).

DETAILED DESCRIPTION:
Lupus erythematosus is an autoimmune disease of unknown origin which is classified according to its clinical features, the course, and laboratory findings. A rough classification divides lupus erythematosus into three subgroups:

1. discoid lupus erythematosus (dLE),
2. subacute cutaneous lupus erythematosus (scLE), and
3. systemic lupus erythematosus (sLEsLE).

The onset of lupus erythematosus affects women three times more frequently than men, with an onset between the 20th and 40th years of life. It is often aggravated or triggered by multiple factors like UV-light, mainly UV-A, hormones (thyroid diseases), pregnancy, oral contraceptives, stress or trauma. Some medications might also play a role as triggering substances, for example antibiotics, psychotropic drugs, beta blockers, procainamide, diuretics, piroxicam, and griseofulvin.

The prevalence of systemic lupus erythematosus (sLEsLE) is 12 to 50/100.000 population worldwide, the incidence is 2 to 8/100.000 per year. Skin disease is one of the most frequent clinical complaints of patients suffering from sLEsLE. It has been found to occur in up to 70% of patients during the course of the disease.

The interesting subgroups of LE that are part of the study population suffer from discoid lupus erythematosus (dLE) or subacute cutaneous lupus erythematosus (scLE) (Fritsch, 1998).

Discoid lupus erythematosus is the most common form of the chronic forms of cutaneous LE. It is a very chronic inflammatory disease consisting of fixed, indurated, erythematous papules and plaques that are often distributed on the head and neck. Without intervention, dLE lesions may last for many years and are associated with extensive scarring. When dLE occurs on the scalp, permanent scarring and alopecia may result. If the initial work-up of a patient with localized lesion of dLE does not reveal evidence of sLEsLE, the risk of developing sLEsLE is low, about 5%. When dLE lesions are generalized, this risk is slightly higher. However, dLE lesions are not uncommon in patients with an established diagnosis of sLEsLE. About 25% of sLEsLE patients will develop lesions of dLE at some time in the course of their disease (Fitzpatrick, 1996).

Subacute cutaneous lupus erythematosus (scLE) was first described in the late 1970s. These patients suffer from cutaneous lesions which have an eruption that is more persistent than that of acute cutaneous lupus erythematosus ("butterfly rash"), lasting weeks to months or longer. The lesions of scLE consist of scaly, superficial, inflammatory macules, patches, papules, and plaques, that are photodistributed, particularly on the upper chest and back, lateral neck, and dorsal arms and forearms. Several different morphologic types of scLE have been described: annular lesions, and two types of papulosquamous lesions, psoriasiform and pityriasiform. About 50% of the patients with scLE will fulfil four or more criteria for the classification of sLEsLE, though most of the scLE patients do not experience serious renal or CNS involvement of lupus erythematosus. Typically, they suffer from skin disease, photosensitivity, and musculoskeletal complaints. Dry eyes and a dry mouth are also not uncommon. Some patients with scLE experience severe manifestations of SLEsLE, and thus all scLE patients should be monitored for systemic disease (Fitzpatrick, 1996).

Frequently, cutaneous complaints are of most concern to patients with scLE and dLE, and thus dermatologists are generally the physicians managing this disease. Broad spectrum sunscreens and sun-protective measures, including lifestyle-changes and clothing are perhaps the most important initial measures. Some patients respond to potent topical steroids. Oral antimalarial therapy is also beneficial in many patients. Less commonly used treatments include dapsone, gold, immunosuppressive drugs, retinoids, and systemic steroids.

Standard treatment with potent topical corticosteroids is very effective but longtime application can provoke atrophy and fragility of the skin as well as telangiectasias erythema perstans, perioral dermatitis and steroid acne. Systemic resorption depending on the dosage, area, and way of application resulting in terms of a dysfunction of the hypothalamus-hypophysis axis has been described (Korting, 1992). Contact allergies are very uncommon, but have been reported (Lauerma et al. 1993).

The main concern is the skin atrophy following long-term application of topical corticosteroids. Therefore the need for alternatives is evident.

Pimecrolimus is an ascomycin and macrolactam derivative, acting as a calcineurin inhibitor which binds calcineurin (Dissemond et al, 2002). The consequence of calcineurin binding is a lack of activation of both T helper cell types 1 and 2. Further effects of these compounds have been suggested on other inflammatory cells, such as Langerhans cells and mast cells/basophils. Both entities, dLE and scLE are characterized by B-cell activation due to affected T-cell activation and the formation of multiple autoantibodies. This results, among other symptoms, in inflammatory infiltrates, especially on the face. Pimecrolimus cream is already approved for the treatment of atopic dermatitis. Furthermore, there have been studies in other indications like psoriasis, allergic and irritant dermatitis. Pimecrolimus has been developed for the potential treatment of psoriasis, allergic, irritant and atopic dermatitis. Animal studies with tacrolimus ointment cream used for lupus dermatoses have shown to be promising (Neckermann et al., 2000; Meingassner et al. 1997; Bochelen et al. 1999). Topical tacrolimus therapy was applied to facial skin lesions in 7 cases of cutaneous lupus erythematosus (cLE). Three systemic LE and one discoid showed a marked regression of their skin lesions after tacrolimus therapy, but three patients with discoid LE were resistant to the therapy. A good response was observed for facial erythematosus lesions with edematous or telangiectatic changes in systemic LE (Yoshimasu et al, 2002, Furukawa et al., 2002). In discoid LE with typical discoid lesions, tacrolimus brought no improvement. Pimecrolimus seems to be more promising than tacrolimus due to the altered skin penetration profile. Topical pimecrolimus cream, in contrast to corticosteroids, does not provoke any skin atrophy (Dissemond et al., 2002; Queille-Roussel et al.; 2001) and might be a good alternative to the standard treatment of potent corticosteroids, even if only a part of the patient population will respond to Elidel® treatment.

Topical formulations of pimecrolimus cream have been shown to be effective in atopic dermatitis, chronic irritant hand dermatitis, allergic contact dermatitis, and also in psoriasis, but in this case, under semi-occlusive conditions. Pharmacokinetic studies with pimecrolimus cream 1% indicate a consistently low systemic exposure in infants, children and adults with atopic dermatitis regardless of the extent of lesions treated and of the duration of therapy. These results support the twice daily administration of pimecrolimus cream in long-term use on an as needed basis, with no limitation on the duration of treatment and on the extent of skin surface area treated. The pimecrolimus cream 1% and the corresponding vehicle were devoid of significant irritation, contact sensitization, phototoxic, or photoallergic potential, in the standard local tolerability studies in healthy volunteers.

The treatment will be without occlusion, since occlusive treatment is not considered clinically relevant for the areas on the face in lupus erythematosus.

Untreated lupus plaques in the same patient show equal expression of the clinical signs of erythema, induration and scaling. This allows the possibility to design a within-patient study to compare the various formulations of interest for efficacy and local tolerability.

Systemic absorption is very low. A pharmacokinetic study of patients with atopic dermatitis who applied 1% pimecrolimus cream twice daily for three weeks did not show any absorption in 72% of the cases. Side effects were not observed (van Leent et al., 1998 a and b).

In view of the biological profile, a clinical hypothesis is formulated claiming that Elidel® is well tolerated and effective in the treatment of cutaneous lupus erythematosus (scLE and dLE). This study is designed to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included only if they fulfil the following inclusion criteria on the pre-treatment days (between Day -14 and Day -2) and on Day 1 (before first application of study medication):

1. Female and male patients aged 18-65 years (females of childbearing potential may be enrolled provided they are routinely using adequate contraception in the assessment of the investigator).
2. Patients with histologically defined dLE or scLE.
3. The test sites (lupus erythematosus plaques) must be on the face only, and have a total sign score of 4 or more (sum of erythema, induration and scaling scores) and must be the same within a given patient (ie not differing in the sum for erythema, induration or scaling). Each of the 2 test sites must be at least 3 cm apart.
4. The patients must receive a baseline medication with chloroquine.
5. Patients must have been informed about the study procedures and medication and must have given their written Informed Consent.
6. Patients expected to be available for the duration of the study and able to comply with the study visits.

Exclusion Criteria:

Any of the following criteria will disqualify a patient from participating in this study:

1. Systemic therapy for lupus erythematosus within one month prior to first application of study medication in this study (steroids, retinoids, herbal medicines, etc) except chloroquine.
2. Patients with systemic lupus erythematosus or patients whose chronic discoid lupus erythematosus appears to be spontaneously flaring or improving based on the experience of the investigator.
3. Patients who are receiving oral medication, known to precipitate lupus lesions (e.g. procainamide, diuretics, piroxicam, beta blockers, griseofulvin, lithium and other psychotropic drugs).
4. Topical therapy [i.e. corticosteroids, etc.] within 2 weeks prior to first application of study medication.
5. Patients with clinically significant medical conditions which could interfere with the conduct of the study. This includes:

   * Renal impairment (creatinine > 2.0 mg/dl)
   * Hepatic impairment (liver function test values above notable abnormalities; g-GT, ALAT, ASAT: 2x the upper limit)
   * Haematologic disorders (haemoglobin, platelet, erythrocyte and leukocyte counts above notable abnormalities)
   * Neurologic disorders (significant impairment of sensory and motor function as judged by the investigator)
   * Patients known to be previously immunocompromised (e.g. lymphoma, AIDS, myelodysplastic disorders) or treated recently with immunosuppressive drugs or treatment (e.g. radiation therapy or chemotherapy). HIV tests are not necessary.
   * Patients with clinically relevant cardio-vascular diseases (New York Heart Association [NYHA] III or IV)
6. Patients who suffer from systemic or generalized infections (bacterial, fungal, viral)
7. Patients with malignancy or history of malignancy.
8. Patients who suffer from acute or chronic bacterial, viral, or fungal skin diseases. However, patients with tinea pedum and/or onychomycosis can be included. Likewise, only patients with acute herpes lesions are excluded.
9. Patients with a history of drug or alcohol abuse during the past 1 year.
10. Patients with known hypersensitivity to any of the ingredients of the study medication or to tacrolimus (the investigator will be provided with a list of ingredients of the study medication).
11. Patients who have received an investigational drug within 4 weeks prior to the first application of the study medication.
12. Patients who are unwilling or unable to provide Informed Consent or to participate satisfactorily for the entire trial period.
13. Any other condition which, in the opinion of the investigator, would render the patient ineligible for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-06

PRIMARY OUTCOMES:
therapeutic effect

SECONDARY OUTCOMES:
local tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sticherling, Prof. Dr. med., Principal Investigator — University of Leipzig, Department of Dermatology
Locations (1):
- Department of Dermatology, University of Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- [Background] Bornhovd EC, Burgdorf WH, Wollenberg A. Immunomodulatory macrolactams for topical treatment of inflammatory skin diseases. Curr Opin Investig Drugs. 2002 May;3(5):708-12. PMID 12090543
- [Background] Katsiari CG, Liossis SN, Dimopoulos AM, Charalambopoulo DV, Mavrikakis M, Sfikakis PP. CD40L overexpression on T cells and monocytes from patients with systemic lupus erythematosus is resistant to calcineurin inhibition. Lupus. 2002;11(6):370-8. doi: 10.1191/0961203302lu211oa. PMID 12139375
- [Background] Wellington K, Jarvis B. Topical pimecrolimus: a review of its clinical potential in the management of atopic dermatitis. Drugs. 2002;62(5):817-40. doi: 10.2165/00003495-200262050-00007. PMID 11929333
- [Background] Eichenfield LF, Lucky AW, Boguniewicz M, Langley RG, Cherill R, Marshall K, Bush C, Graeber M. Safety and efficacy of pimecrolimus (ASM 981) cream 1% in the treatment of mild and moderate atopic dermatitis in children and adolescents. J Am Acad Dermatol. 2002 Apr;46(4):495-504. doi: 10.1067/mjd.2002.122187. PMID 11907497